CLINICAL TRIAL: NCT02792361
Title: A Randomized, Non-Blind, Clinical Effectiveness Trial in Post-Operative Pterional Craniotomy Drain Placement
Brief Title: A Clinical Effectiveness Trial in Post-Operative Pterional Craniotomy Drain Placement
Acronym: EPOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Wyatt Ramey, Medical Doctor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SCT1121
Record Dates: First submitted 2016-05-25; First posted 2016-06-07 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-05

CONDITIONS: Pterional Craniotomy
Keywords: Post-Operative Pterional Craniotomy; Suction Drain; Benefits

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Subjects who did not have a suction drain placed post-operatively following a Pterional Craniotomy.
- Treatment Group (Experimental): Subjects who did have a suction drain placed post-operatively following a Pterional Craniotomy at the location of surgical incision.
  Interventions: Procedure: Standard Suction Drain

INTERVENTIONS:
Procedure: Standard Suction Drain — The intervention of the experimental group will be a standard suction drain placed at the surgical site following a Pterional Craniotomy.
  Arms: Treatment Group

SUMMARY:
This is a clinical trial where patients who present to the neurosurgery service in need of a procedure that requires a pterional craniotomy will be screened, and if eligible, enrolled for the randomization in the placement of a drain at the surgical site. At present, there is not a protocol for whether or not to use a drain following this procedure. There is some debate on whether it serves any real benefit for the patient or if it may actually be detrimental in cases where infection occurs. This study aims to answer this question by randomizing patients to drain placement and then comparing patient outcomes between the two groups. These include the following: infection rate, length of hospital stay, self-reported patient pain and discomfort, the amount of time before patients are able to open their eye ipsilateral to the side of operation, change in forehead circumference post-op days 1-3, and any unforeseen post-operative complications. This will be accomplished through using a patient-administered survey, recording physical measurements, and a patient chart review. Statistical analysis will then be used to identify any differences that may exist.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have been scheduled for surgery requiring the use of a pterional craniotomy approach

Exclusion Criteria:

* Patients in need of a surgical intervention requiring a pterional craniotomy due to reasons of physical injury
* Patients who need a pterional craniotomy with a orbitozygomatic approach
* Patients who have noticeable physical injury to their skull
* Patients with a prior surgical history of a craniotomy
* Patients with a pathological condition deemed severe enough by the screening physician to possibly influence the healing process of the procedure (blood clot disorder, cirrhosis, severe nutrient depletion, congestive heart failure etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Difference in Length of Hospital Stay | From the date of surgery to the date of discharge from the hospital for up to 16 weeks following surgery, or until death, depending which comes first.
  Compare the length of hospital between the treatment groups and determine whether a significant difference exists.
Head Circumference Difference | Day 1 through Day 3 following surgery.
  Compare the change in measured forehead circumference between treatment groups on post-operative days 1-3. Determine if a significant difference exists between the two.
Pain Difference | At the time of discharge from the hospital but no longer than up to 16 weeks from the date of surgery.
  Compare the reported pain/ discomfort between the patients who had drain placement from those who did not. This will be performed using a survey administered to patients upon removal of the drain
Ability to open ipsilateral eye to surgical site. | Day 1 through Day 3 following surgery.
  Compare the number of subjects able to open and close their eye on the ipsilateral side of the surgical site between the study groups
Complication Rate | From the date of surgery to the date of discharge from the hospital for up to 16 weeks following surgery, or until death, depending which comes first.
  An overall assessment comparing complications between the two study groups will be performed. This will include looking things such as hospital acquired pneumonia, the development of any new neurological conditions or deficiencies, and other unforeseen complications that may arise which are not be directly related to the drain but may potentially still be influenced by it.
Surgical site infection rate | From the date of surgery to the date of discharge from the hospital for up to 16 weeks following surgery, or until death, depending which comes first.
  Compare infections rates between patients with drains placement versus those who did not. Determine if there is any statistically significant difference in risk exists between the two study populations.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available. However, findings may be published in a peer-reviewed academic journal.

REFERENCES:
- [Background] Chaddad-Neto F, Campos Filho JM, Doria-Netto HL, Faria MH, Ribas GC, Oliveira E. The pterional craniotomy: tips and tricks. Arq Neuropsiquiatr. 2012 Sep;70(9):727-32. doi: 10.1590/s0004-282x2012000900015. PMID 22990732
- [Background] Dougherty SH, Simmons RL. The biology and practice of surgical drains. Part II. Curr Probl Surg. 1992 Sep;29(9):633-730. doi: 10.1016/0011-3840(92)90028-2. No abstract available. PMID 1424760
- [Background] Cruse PJ, Foord R. A five-year prospective study of 23,649 surgical wounds. Arch Surg. 1973 Aug;107(2):206-10. doi: 10.1001/archsurg.1973.01350200078018. No abstract available. PMID 4719566
- [Background] Mollman HD, Haines SJ. Risk factors for postoperative neurosurgical wound infection. A case-control study. J Neurosurg. 1986 Jun;64(6):902-6. doi: 10.3171/jns.1986.64.6.0902. PMID 3701440